CLINICAL TRIAL: NCT03135002
Title: The Leicester City and County Chronic Kidney Disease Study: An Observational Chronic Kidney Disease Cohort to Study Cardiovascular and Renal Outcomes in Multi-ethnicity Primary Care
Brief Title: The Leicester City and County Chronic Kidney Disease Cohort
Acronym: LCC-CKD
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); Leicester City Clinical Commissioning Group (Unknown); West Leicestershire Clinical Commissioning Group (Unknown); East Leicestershire Clinical Commissioning Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0576
Record Dates: First submitted 2017-04-19; First posted 2017-05-01 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-05

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Other

SUMMARY:
Chronic kidney disease (CKD) is estimated to affect 6-8% of the adult population and is independently associated with increased cardiovascular (CV) disease risk. This risk increases as CKD advances both in relation to worsening glomerular filtration rate and development of proteinuria. The overall cost of CKD to the NHS (National Health Service) in England has been estimated as £1.45 billion per annum, or 1.3% of the NHS's total budget. This includes £175 million, or 13% of the CKD budget, annually spent in relation to 19,000 excess myocardial infarctions and strokes related to CKD.

The epidemiology of CKD in primary care is poorly studied. This is particularly the case in non-white populations who have an independent higher risk of progression to end stage renal failure (requiring dialysis or transplantation), CV events and death.

Further, CV disease risk in CKD remains poorly described beyond simple risk stratification by CKD stage. A recent systematic review identified some CKD-specific CV disease risk scores. However, all the risk scores had significant methodological limitations, such as a lack of external validation or the perception that they were not 'clinically useful'. The Leicester City and County Chronic Kidney Disease (LCC-CKD) cohort will be created from anonymised GP (general practice) records of individuals with CKD. We will aim to retrospectively create a cohort with 5 years follow-up to the present day. In addition, a present day cohort will be created to both aid research and provide data for practices and clinical commissioning groups for quality improvement (QI) purposes. We will aim to include 30,000 individuals with CKD in the cohort.

The principal objectives of the study are:

1. To study the natural history of CKD in a multi-ethnic primary care setting
2. To contribute to the creation of a risk prediction tool for heart attacks and strokes in CKD

The risk prediction tool would more accurately stratify risk of CV events for individuals with CKD. This would aid patients and clinicians in deciding on treatments aimed at reducing the risk of future myocardial infarctions and strokes. Currently, individuals with CKD, despite higher risk of CV disease, may not be receiving optimum treatment such as statins and anti-hypertensive medications. Improved management of cardiovascular risk factors in CKD is likely to see a reduction in CKD associated excess CV events and their associated costs, including longer average duration of inpatient admissions.

ELIGIBILITY:
Inclusion Criteria:

* Practice Level - all primary care practices within the 3 Clinical Commissioning Groups participating in the study.
* Patient Level - any individual 18 years or over with an MDRD (Modification of Diet in Renal Disease) or CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) eGFR (estimated glomerular filtration rate) less than 60ml/minute/1.73m2, proteinuria or a Read code CKD diagnosis.

Exclusion Criteria:

* Aged less than 18 years of age
* Endstage renal failure i.e. already receiving dialysis or with a kidney transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with non-endstage chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease events | 5 years
  Major cardiovascular events, to study the natural history of CKD in a multi-ethic primary care setting and to contribute to the creation of a risk prediction tool for heart attacks and strokes in CKD

SECONDARY OUTCOMES:
All-cause mortality | 5 years
Hospitalisation | 5 years
  For individuals with CKD is associated with increased length of stay and therefore cost

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided